CLINICAL TRIAL: NCT02676037
Title: Diagnosis of Hallux Valgus by Using a Foot Pressure Platform as an Alternative to Radiological Images
Status: Completed | Type: Observational
Sponsor: University of Dundee (Other)
Responsible Party: Principal Investigator, Rami Abboud, Director of Institute of Motion Analysis and Research, University of Dundee
Other Study IDs: 2015OS06
Record Dates: First submitted 2016-02-02; First posted 2016-02-05 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Hallux Valgus
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 9 Months

INTERVENTIONS:
Device: foot pressure plate form

SUMMARY:
Hallux Vagus is a common deformity which affects the first metatarsalphalangeal joint. The current diagnostic tool is using X-ray which is expensive and includes radiation exposure. The current study is aimed at using the foot pressure platform as an alternative method for diagnosis and evaluation of the deformity. The main subjects will be recruited from orthopaedic outpatient clinics.

The recruited subjects will undergo the non-invasive and radiation free study by walking on a pressure platform. Then their pressure data will be correlated with their radiological study which has already been done in the clinic. The aimed outcome of the study is use the foot pressure platform as first line of diagnosis and evaluation of the Hallux Valgus deformity.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with hallux valgus.
* Patients who are diagnosed with hallux valgus and scheduled for surgery ( to be seen pre and post-surgery)
* Patient who are diagnosed with hallux valgus and had surgery

Exclusion Criteria:

* Any other foot deformity
* Previous foot surgery (which is not related to HV

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will come from an existing list of patients referred to the Foot Pressure Analysis Clinic and will include any patients who are diagnosed with HV. They will be recruited with the knowledge of the consultant orthopedic surgeons who are the direct care providers for these patients. The surgeons will write to eligible participants and include a Patient Information sheet about the project (which does not require to record data beyond what is normally performed as part of the Foot Pressure Analysis Clinic) If the participant is interested in taking part he/she will contact the department.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
- To provide a safe diagnostic tool (radiation free) for evaluating the severity of the HV by using a foot pressure platform | 2 years

IPD SHARING:
Plan to Share IPD: Undecided